CLINICAL TRIAL: NCT07109999
Title: Biomarker-based Alzheimer's Disease Cohort Study (BASIC)
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2024347
Record Dates: First submitted 2025-05-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with Alzheimer's disease with AD biomarker positivity.: This cohort recruits patients diagnosed with Alzheimer's disease based on clinical symptoms, neuroimaging features and AD biomarkers. Biomarker positivity is necessary for inclusion.
  Interventions: Other: None-placebo

INTERVENTIONS:
Other: None-placebo — This study is an observational study, and no interventions will be implemented.

SUMMARY:
This study adopts a prospective cohort design, constructing a single-center cohort by recruiting patients with Alzheimer's disease (AD) who are positive for AD biomarkers. First, the investigators aim to establish a cohort of AD patients with positive biomarkers, thereby reserving suitable patient resources for future AD-related clinical trials. Second, based on the established cohort, the investigators will explore the associations between AD-related biomarkers and clinical manifestations among the elderly population in China, and identify potential risk factors influencing the progression of AD. Third, according to the identified risk factors for AD progression, the investigators will construct a risk early warning model for the progression rate of AD based on biomarkers, in order to achieve early identification and precise prevention and control of the progression risk of AD.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients aged 40 years or older;
* (2) Visiting Xuanwu Hospital, Capital Medical University;
* (3) Meeting the core clinical diagnostic criteria for Alzheimer's disease (AD) - related mild cognitive impairment or probable AD according to the NIA-AA (2011);
* (4) Amyloid positivity confirmed by amyloid PET or cerebrospinal fluid biomarker tests;
* (5) Providing informed consent.

Exclusion Criteria:

* (1) Individuals who are unable to complete the assessment due to severe psychological or physiological disorders.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls individuals aged 40 years or older who are under evaluation or care at Xuanwu Hospital, Capital Medical University. Eligible participants must meet the National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical diagnostic criteria (2011) for Alzheimer's disease (AD)-related mild cognitive impairment or probable AD. All included individuals are required to demonstrate amyloid positivity via validated biomarker testing, such as amyloid positron emission tomography (PET) imaging or cerebrospinal fluid analysis. Participants must also provide written informed consent to participate in the study. Individuals with severe psychiatric or neurological conditions that would preclude their ability to complete standardized assessments or comply with study protocols are excluded from enrollment. This cohort aims to characterize a clinically and biomarker-confirmed AD population for research on disease progression or therapeutic interventions.
Sampling Method: Non-Probability Sample
Enrollment: 2835 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
The event of conversion from mild cognitive impairment to dementia within three years. | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The event of conversion from mild cognitive impairment to dementia within three years. Cognitive status will be assessed using Clinical Dementia Rating scale-Global Score (CDR-GS): mild cognitive impairment: CDR-GS = 0.5; dementia: CDR-GS > 0.5.

SECONDARY OUTCOMES:
Hachinski Ischemia Score | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The Hachinski Ischemic Score (HIS) is a brief 13-item scale (range 0-18) in which scores ≤4 favor Alzheimer's disease and ≥7 suggest vascular dementia, based on clinical features such as abrupt onset, vascular risk factors, and focal neurological signs.
Memory - Immediate Recall | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Immediate Recall assesses short-term auditory-verbal memory by recording the number of words correctly repeated after a single presentation (typically 0-15); lower scores indicate poorer encoding.
Digit Span Test | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Digit Span Test quantifies auditory-verbal working memory via the longest sequence of digits correctly repeated forward (attention) and backward (manipulation); score = maximum span length.
Trail Making Test (TMT) | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Trail Making Test (TMT) measures processing speed and executive function via completion time (seconds) for Part A (number sequencing) and Part B (alternating numbers-letters); higher scores indicate poorer performance.
Boston Naming Test | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Boston Naming Test quantifies confrontation naming ability by the number of spontaneously correct responses; lower scores indicate lexical-semantic impairment.
Memory - Delayed Recall | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Delayed Recall quantifies the number of previously learned items correctly reproduced after a ≥20-minute unfilled interval (range 0-15); lower scores signal impaired consolidation.
Memory - Cued Recall | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Cued Recall evaluates the number of previously learned items correctly retrieved following semantic prompts (range 0-15); lower scores reflect deficient retrieval efficiency.
Subjective Cooperation Score | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Subjective Cooperation Score is a single-item rater judgment (0-10 scale) quantifying participant engagement and compliance during cognitive testing; higher values denote greater cooperation.
Neuropsychiatric Inventory (NPI) | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The Neuropsychiatric Inventory (NPI) is a validated informant-based scale assessing 12 neuropsychiatric domains (range 0-144); higher scores denote greater symptom frequency and severity.
Geriatric Depression Scale (GDS) | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The 15-item Geriatric Depression Scale (GDS-15) is a self-report screen for depressive symptoms in older adults; total score 0-15, with ≥5 indicating probable depression.
Daily and Overall Functional Assessment | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Daily and Overall Functional Assessment quantifies independence in basic and instrumental activities of daily living (ADL/IADL) via standardized informant or performance-based scales; higher scores denote greater functional ability.
Activities of Daily Living (ADL) | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The Activities of Daily Living (ADL) Scale is a brief, validated instrument that rates independence in basic self-care tasks; scores range from 0 (total dependence) to 6 (full independence), with lower values indicating greater functional impairment.
Clinical events | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  The events of transitioning from mild dementia to moderate dementia, and from moderate dementia to severe dementia.Cognitive status will be assessed using Clinical Dementia Rating scale-Global Score (CDR-GS): mild cognitive impairment: CDR-GS = 0.5; moderate dementia: CDR-GS = 2; severe dementia: CDR-GS = 3.
Blood biomarkers | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Amyloid-beta (Aβ), tau, neurofilament light chain protein (NFL), brain-derived neurotrophic factor (BDNF), glial fibrillary acidic protein (GFAP), and markers related to chronic inflammation, etc.
Magnetic resonance imaging (MRI) examination | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Structural imaging and functional imaging.
Electroencephalogram (EEG) | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Power of each EEG frequency band
Polysomnography | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
Positron Emission Tomography (PET) scan | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Brain metabolic imaging and amyloid imaging
Cerebrospinal fluid (CSF) examination | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.
  Routine and biochemical analysis of cerebrospinal fluid (CSF), as well as the measurement of Aβ and tau proteins
Near-infrared brain functional imaging | Assessments will be conducted every 6 months to 1 year upto 15 years for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China